CLINICAL TRIAL: NCT03895294
Title: Effect of Strategic Purchasing of Antiviral Drugs and the Clinical Pathway for the Treatment of Chronic Hepatitis C in Colombia
Brief Title: Effect of Strategies for the Treatment of Chronic Hepatitis C in Colombia
Acronym: HEPCSTRATEGY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Universidad de Antioquia
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis C
Keywords: Direct-Acting Antivirals; Health Services Accessibility
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health care under the strategic purchase-Clinical pathway (Experimental): Health care under the strategic purchase and the Clinical pathway for the treatment of chronic Hepatitis C
  Interventions: Other: Health care under the strategic purchase-Clinical pathway
- Usual care process prior strategic purchase-clinical pathway (Active Comparator): Usual care process prior to the establishment of the strategic purchase and the Clinical Pathway
  Interventions: Other: Usual care process prior strategic purchase-clinical pathway

INTERVENTIONS:
Other: Health care under the strategic purchase-Clinical pathway — 1) purchase of DAA by the MoHSP; 2) diagnosis of the patient (confirmed by quantitative HCV RNA test); 2) prescription of the treatment by a specialist in internal medicine, hepatology or Infectious disease; 3) daily supervised drug administration by a nurse or weekly treatment dispensing by pharmacist; 4) Pharmaceutical Care (includes: consultation with pharmacist at weeks 0, 4, week of the end of treatment (8, 12 or 24) and week of evaluation of effectiveness (week 12 or 24 after the end of treatment); health education and administrative support. In case of identifying any Drug-related Problem, the respective pharmaceutical intervention was made.
  Arms: Health care under the strategic purchase-Clinical pathway
Other: Usual care process prior strategic purchase-clinical pathway — 1) diagnosis of the patient (confirmed by quantitative HCV RNA test); 2) prescription of the treatment by a specialist in hepatology; 3) weekly treatment dispensing by pharmacist; 4) patient use; 5) Pharmaceutical Care (includes: consultation with pharmacist at weeks 0, 4, 8, week of the end of treatment (12 or 24) and week of evaluation of effectiveness (week 12 or 24 after the end of treatment); health education and administrative support). In case of identifying any Drug-related problem, the respective pharmaceutical intervention was made.
  Arms: Usual care process prior strategic purchase-clinical pathway

SUMMARY:
Hepatitis C is a public health problem and the high cost of the Direct-Acting Antivirals (DAA) is one of the main limitations for treatment worldwide.

In Colombia, the Ministry of Health and Social Protection (MoHSP) has made progress in addressing Hepatitis C problem in order to control the infection and resolve barriers to access to medicines. One of the strategies implemented was the purchase of DAA, in association with the PAHO, and the instauration of the Clinical Pathway for the treatment of chronic hepatitis C.

The implementation of the Clinical Pathway has required the integration of health care processes and the respective report in the health information systems, allowing a high level of control in the monitoring of the Hepatitis C and the subsequent generation of indicators. However, there is limited information on the effects of the strategic purchase and the instauration of the Clinical Pathway on the costs of care, clinical outcomes and the quality of health care for patients with Hepatitis C in Colombia.

The aim of this study is to establish the effect of strategic purchasing and the Clinical Pathway for the treatment of chronic Hepatitis C, in the clinical results, in the general costs and quality of health care of Hepatitis C patients in Colombia.

DETAILED DESCRIPTION:
A quasi-experimental design with a non-equivalent control group will be performed, where there will be an intervention group and a control group formed naturally before the investigation. In order to reduce the possible selection bias due to the lack of randomization, the propensity score method will be used. 62 patients will be included in each arm.

An estimation and comparison of the direct costs of the care of patients with Hepatitis C, before and after the implementation of the strategic purchase and the Clinical Pathway will be made, using a "top to bottom" method.

A questionnaire will be applied to the patients of the intervention group in order to identify barriers and facilitators to Hepatitis C health care and patient satisfaction with health care process under the Clinical Pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Chronic Hepatitis C confirmed by quantitative HCV RNA test
* Patient affiliated to the contributory system of one Health Promoting Enterprise from Colombia.
* Patients with prescription of pharmacological treatment for Hepatitis C.

Exclusion Criteria:

* Patients with incomplete information in at least one of the following variables: fibrosis, cirrhosis (if applicable), antiviral drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Access to treatment | 2 months
  Proportion of patients who initiates treatment, in comparison with the total number of patients with indication of treatment (confirmed diagnosis and prescription of treatment).

SECONDARY OUTCOMES:
Opportunity at the start of treatment | 2 months
  The difference in days between the date of the first prescription of the antiviral treatment and the start date.
Effectiveness | 6 months
  Proportion of treated patients that achieved Sustained Virological Response (SVR), that is, undetectable HCV viral load (lower than the Lower Quantification Limit -LL-), 12 weeks after the end of the DAA therapy (SVR12) or 24 weeks after the end of treatment for the schemes that include interferon (SVR24)
Drug-related problem | 6 months
  Proportion of patients who initiated treatment and who presented at least one Drug-Related Problem registered in the clinical history, database and / or pharmacovigilance reports.

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Ledezma, Msc, Principal Investigator — Universidad de Antioquia; Pedro Amariles, PhD, Study Director — Universidad de Antioquia; Andrea Salazar, PhD, Study Chair — Universidad de Antioquia
Locations (1):
- Medicarte, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical pathway for the treatment of chronic Hepatitis C, a look and a complement from the perspective of pharmaceutical services — http://www.scielo.org.co/scielo.php?script=sci_arttext&pid=S0120-99572018000400483